CLINICAL TRIAL: NCT03964285
Title: Impact of Rumination on Affectivity After Physical Activity in Fibromyalgia
Brief Title: Repetitive Thinking in Fibromyalgia
Acronym: PRFM-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Université de Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2018_843_0035
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rumination; Fibromyalgia; Chronic Pain; Repetitive Negative Thinking
Keywords: Rumination; Fibromyalgia; Chronic Pain; affectivity; repetitive negative thinking
MeSH Terms: conditions — Rumination Syndrome; Fibromyalgia; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rumination group (Active Comparator): The patients will receive rumination induction. Rumination induction will follow a relevant activity for our patients: climbing steps. Rumination induction will be done right after climbing the steps.
  Interventions: Other: rumination induction
- distraction group (Experimental): Distraction will follow a relevant activity for our patients: climbing steps. Distraction induction will be done right after climbing the steps.
  Interventions: Other: distraction induction

INTERVENTIONS:
Other: rumination induction — The induction method is based on specific instructions given to participants on how to focus on different elements of their experience. For example, they will be led, in the rumination condition, to reflect on the causes, meanings and consequences of the amount of tension they feel in their muscles.
  Arms: Rumination group
Other: distraction induction — The induction method is based on specific instructions given to participants on how to focus on different elements of their experience. In the distraction condition they will, for example, imagine a ship crossing the Atlantic.
  Arms: distraction group

SUMMARY:
Some fibromyalgia patients may use inappropriate emotional regulation strategies to respond to pain. Rumination could be one of this inefficient regulation strategies. The investigators believe that the use of rumination strategies to respond to the discomfort of daily physical activity would maintain and aggravate a negative emotional state after the effort. Distraction would be a more effective strategy to cope with pain. From this data, the investigators want to explore the causal link between rumination and negative affectivity after physical activity in fibromyalgia using an experimental design.

DETAILED DESCRIPTION:
Fibromyalgia is a disorder characterized by widespread musculoskeletal pain accompanied by fatigue, sleep, memory and mood issues. As with any condition of chronic pain, psychological mechanisms can help maintain discomfort and pain. These mechanisms may hinder the recovery of physical activity. Some patients may use cognitive strategies of emotional regulation that are ineffective to cope with pain and discomfort of everyday activities, such as rumination. The literature suggests that this process is linked to the physical and psychological difficulties of fibromyalgia. However, no study has revealed a causal link between rumination and negative affectivity in a context of physical activity in this population. The investigators want to test this hypothesis by directly manipulating the style of information processing following a relevant activity for these patients: climbing steps. In one group the investigators will induce rumination right after climbing the steps. In the other group the investigators will induce distraction. Patient with Fibromyalgia will be recruited at the Pain Center of CHU-Amiens. Patients will complete different scales before to climb steps and after experimental induction. The investigators hypothesize that Patients using a rumination strategy after an uncomfortable physical activity will experience a greater subjective discomfort than patients using a distraction strategy.

ELIGIBILITY:
Inclusion Criteria:

* Adults Patients
* Free and informed consent signed.
* French native speaker, writer and reader.
* according 1990 American College of Rheumatology criteria : Patients with diffuse pain for more than three months and with digital palpation pain on more than 11 insertion points.

Exclusion Criteria:

* minor patients
* Adult major under administrative protection
* Patient with severe psychosis or depression or severe anxiety or impulsivity as assessed by the clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change in PANAS score before and after induction phase | One hour and twenty minutes after inclusion of the patients
  The PANAS Scale or Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire. The list is split up into two segments, or mood scales. One scale measures a person's positive emotion and the other scale measures the negative. Each segment has ten terms, which can be rated on a scale of 1 to 5 to indicate the extent to which the respondent agrees that this applies to him.Characteristic of this test is the fact that it can be completed in 10 minutes. High score is associated with stress and anxiety. small score is associated with calm.

SECONDARY OUTCOMES:
Change in VAS score before and after induction phase | One hour and twenty minutes after inclusion of the patients
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions. The patient is asked to place a vertical mark on the scale to indicate the level of intensity of his or her pain, anxiety, depression, etc. 0 would mean "no pain" and 10 would mean "worst possible pain."

CONTACTS AND LOCATIONS:
Overall Officials: Eric Serra, MD, Principal Investigator — CHU Amiens; Virginie Marechal, MD, Principal Investigator — CHU Amiens; Alain DERVAUX, MD, Principal Investigator — CHU Amiens; Jérémy Fonseca Das Neves, PhD, Principal Investigator — CHU Amiens; Stéphane Rusinek, PHD, Principal Investigator — Lille University
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fonseca das Neves J, Kornacka M, Serra E, Rollin N, Kosinski T, Marechal V, Jehel L, Rusinek S. The impact of rumination on fibromyalgia pain after physical activity: an experimental study. Sci Rep. 2023 Nov 22;13(1):20523. doi: 10.1038/s41598-023-47414-z. PMID 37993555